CLINICAL TRIAL: NCT01113827
Title: Effects of Water-soluble Olive Extract on Antioxidant Status, Exercise Performance, Muscle Metabolism, Muscle Damage and Inflammation
Brief Title: Effects of Water-soluble Olive Extract Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2009-09-01-OLIV
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Olive; antioxidant; exercise; inflammation; recovery; Healthy men
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — olive extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 150mg olive extract (Active Comparator)
  Interventions: Dietary Supplement: Olive Extract
- 50mg olive extract (Active Comparator)
  Interventions: Dietary Supplement: Olive Extract
- Placebo control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Olive Extract — Capsule form ingested 1x/day for 6 weeks
  Arms: 150mg olive extract; 50mg olive extract
Dietary Supplement: Placebo — Placebo
  Arms: Placebo control

SUMMARY:
Six weeks of supplementation of an olive extract will:

* Improve antioxidant status
* Reduce inflammation
* Reduce muscle damage
* Improve exercise performance
* Improve exercise recovery as compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Recreational exerciser
* BMI <= 30
* Non-smoker

Exclusion Criteria:

* Blood pressure over 140/90
* Type I or Type II diabetes
* Renal, hepatic or cardiac disease
* Current infectious disease

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Improved Antioxidant Status | 6 weeks

SECONDARY OUTCOMES:
Reduced Inflammation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Ivy, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States